CLINICAL TRIAL: NCT02574195
Title: Evolution of Effectiveness of Diabetes Medical Care in Russia
Status: Completed | Type: Observational
Sponsor: Endocrinology Research Centre, Moscow (Other Government)
Responsible Party: Sponsor
Other Study IDs: ESR1410209
Record Dates: First submitted 2014-12-18; First posted 2015-10-12 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus; microvascular complications; macrovascular complications; epidemiology; Russia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The main aim of the present study is to evaluate the prevalence of individual microvascular and macrovascular complications among diabetes mellitus patients and to determine the percentage of diabetes mellitus patients achieved HbA1c<7,0%.

DETAILED DESCRIPTION:
Rationale for this Study Primary Existing routine health statistics underestimates the rate of morbidity due to diabetes complications. To provide more realistic estimation of morbidity, repeated epidemiological studies are essential in assessment of tendencies in diabetes medical care at the country level. They allow to reveal issues, which, being resolved, can contribute to the improvement of diabetes medical care effectiveness. Guidelines developed with this study data may save healthcare budgets and prevent financial losses due to diabetes-related morbidity and disability.

Objectives of the Study • Primary objective: To determine the prevalence of individual microvascular and macrovascular complications among patients with diabetes mellitus type 1 and type 2

• Secondary objective: To determine the percentage of patients with diabetes mellitus type 1 and type 2 achieved HbA1c <7,0%.

Study design The hired medical team (9 specialists) is going to perform the technical study-related tasks in Moscow Region.

Target population includes approximately 147,000 diabetes mellitus patients included in Regional Diabetes Mellitus Register, from which patients will be selected via random sampling (600 patients).

A special rented medical bus will accommodate the study personnel at the place and all the local study-related activities.

After obtaining a written Informed Consent Form by local endocrinologist the each study subject will have one study visit, when he or she should appear fasting and the following data will be collected, tests and examination performed:

* date of the diagnosis of type 1 or type 2 diabetes mellitus;
* medical history including coronary heart disease, myocardial infarction, coronary revascularization, cerebrovascular disease (ischaemic stroke, a transient ischemic attack), peripheral artery disease, diabetic retinopathy (type, stage, year of diagnosis), diabetic neuropathy, chronic kidney disease, diabetic foot;
* blood tests for HbA1c, serum total cholesterol, triglycerides, HDL- cholesterol, serum creatinine and estimation estimated Glomerular filtration rate by standard CKD-EPI, alanine-aminotransferase, aspartate-aminotransferase;
* urine analysis for albumin in spot urine;
* measurement of height, weight/BMI;
* measurement of sitting blood pressure, Electocardiogramm;
* eye examination, including fundoscopy;
* foot examination, including tests for touch, pain, temperature, and vibration sensation of the toes and mini-doppler ultrasound vessel study;
* current pharmacological therapy regimen (medications, daily doses). The medical team will admit up to 35 study subjects per day. This study has descriptive character. There is no any comparison to be performed.

ELIGIBILITY:
Inclusion criteria:

The subject population for this study must meet the following criteria:

1. Provision of singed subject informed consent
2. Type 1 and type 2 diabetes mellitus Target population includes approximately 147,000 diabetes mellitus patients included in Regional DM Register, from which patients will be selected via random sampling (600 patients).

The prescription of the medicinal product is clearly separated from the decision to include the subject in the study.

Exclusion criteria:

1. Diagnosis of gestational diabetes mellitus alone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 or type 2 Diabetes Mellitus
Sampling Method: Non-Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with diabetes mellitus type 1 and type 2diabetes mellitus complications | 30 days
  macrovascular complications, i.e. with history of
  * chronic heart disease
  * myocardial infarction
  * ischaemic stroke
  * transient ischemic attack
  * any revascularization procedure
  * any peripheral atherosclerosis
    e) microvascular complications, i.e.
  * diabetic retinopathy
  * diabetic neuropathy
  * albuminuria
  * chronic kidney disease stage f) other complications diagnosed after diabetes mellitus has been established, i.e.
  * foot examination findings

SECONDARY OUTCOMES:
The percentage of patients with diabetes mellitus type 1 and type 2 achieved HbA1c <7% | 30 days
Structure of antidiabetic therapy (% insulin, % OAD mono, % OAD dual, % OAD triple) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Marina Shestakova, Principal Investigator — ERC Moscow
Locations (1):
- Endocrinology Scientific Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided